CLINICAL TRIAL: NCT00561119
Title: Phase III, Multicenter, Randomized Trial of Maintenance Versus Observation After Achieving Clinical Response in Pts With Metastatic or Recurrent Breast Cancer Who Received 6 Cycles of Gemcitabine Plus Paclitaxel(GP) as 1st-line Chemotherapy
Brief Title: Maintenance Versus Observation After 6 Cycles of Gemcitabine Plus Paclitaxel in Pts With Advanced Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: Korean Cancer Study Group (Other)
Responsible Party: Principal Investigator, Young-Hyuck Im, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007-03-003
Record Dates: First submitted 2007-11-18; First posted 2007-11-20 (Estimated); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: Advanced Breast Cancer
Keywords: maintenance chemotherapy; metastatic or recurrent breast cancer; gemcitabine; paclitaxel(GP)
MeSH Terms: conditions — Neoplasm Metastasis; Breast Neoplasms | interventions — Gemcitabine; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (No Intervention): Observation after 6 cycles of gemcitabine plus paclitaxel till progression
- Arm 2 (Experimental): Maintenance chemotherapy with gemcitabine plus paclitaxel after 6 cycles of gemcitabine plus paclitaxel till progression
  Interventions: Drug: gemcitabine , paclitaxel

INTERVENTIONS:
Drug: gemcitabine , paclitaxel — Gemcitabine 1250 mg/m2 i.v. Day 1 & 8
  Paclitaxel 175 mg/m2 i.v. day 1
  repeat every 3 weeks
  Arms: Arm 2

SUMMARY:
The primary goal of therapy in patients with metastatic breast cancer is palliation and prolongation of life with quality. Although there are no randomized trials comparing chemotherapy with supportive care in women with metastatic breast cancer, chemotherapy clearly provides a survival benefit in metastatic breast cancer. Due to diagnosis at earlier phases of metastatic disease and more effective therapies, the median survival of patients treated with modern taxane-based chemotherapy is now reaching approximately 2 years. The duration of chemotherapy in patients responding or stable disease remains controversial, since quality of life is not usually adversely affected and may even be improved in many patients receiving cytotoxic chemotherapy. In addition, many commonly used chemotherapeutic agents are not limited by cumulative toxicity in metastatic breast cancer patients. Several studies investigated the role of maintenance chemotherapy suggest that maintenance chemotherapy is associated with superior time to progression but no survival gain. However, these randomized trials did not incorporate taxane-based chemotherapeutic regimens, the new standard of care in metastatic breast cancer patients these days. A 1998 metaanalysis of 1,986 patients randomly assigned between combination chemotherapy and single-agent therapy in metastatic breast cancer patients demonstrated a survival advantage to combination chemotherapy, with a hazard ratio of 0.82 (range, 0.75 to 0.90). Although there are several randomized trials showing negative results for survival gain in patients who received maintenance chemotherapy, the role of maintenance chemotherapy with newer agents, such as docetaxel or paclitaxel, have not been established yet. Although Italian MANTA trial demonstrated no difference in PFS or survival between the two arms, their metaanalysis advocated survival benefit of maintenance therapy. Since gemcitabine/paclitaxel (GP) combination chemotherapy is one of the two regimens which showed definite survival gain with favorable toxicity from a randomized trial, we plan to randomize patients who responded to six cycles of GP induction chemotherapy to receive additional maintenance GP chemotherapy until disease progression versus observation. We hypothesize that patients who receive maintenance GP chemotherapy will do better in terms of progression free survival.

DETAILED DESCRIPTION:
The primary goal of therapy in patients with metastatic breast cancer is palliation and prolongation of life with quality, because many if not most patients with metastatic breast cancer ultimately die of their disease. Although there are no randomized trials comparing chemotherapy with supportive care in women with metastatic breast cancer, chemotherapy clearly provides a survival benefit in early breast cancer and produces tumor shrinkage in metastatic disease. Institutional databases show an improvement in the survival of patients with metastatic disease over the past two decades, which may be due to diagnosis at earlier phases of metastatic disease and more effective therapies. The median survival of patients treated with modern taxane-based chemotherapy is now reaching approximately 2 years.

The duration of chemotherapy in patients responding or stable disease remains controversial, since quality of life is not usually adversely affected and may even be improved in many patients receiving cytotoxic chemotherapy. In addition, many commonly used chemotherapeutic agents are not limited by cumulative toxicity in metastatic breast cancer patients. Several trials have reported that continuous therapy generally prolonged the duration of remission, but the effect on survival and quality of life were less consistent.

Coates et al compared continuous therapy with AC or CMF with intermittent therapy using 3 cycles of the same regimen with reinstitution of therapy at the time of disease progression. Patients receiving continuous therapy had superior response rates, time to progression, and better quality of life, but no improvement in overall survival in this trial. A similar trial by the Peidmont Oncology Association randomly assigned patients who had responding or stable disease after six cycles of CAF to either CMF or observation, followed by reinstitution of CMF at disease progression . Although time to progression was more than twice as long for patients on continuous therapy than for those with interrupted treatment, overall survival was similar. Falkson et al randomly assigned 141 patients whose measurable disease showed a complete response after 6 cycles of CAF to receive either chemohormonal therapy or observation and found no difference in overall survival despite of prolongation of time to progression in treatment arm . In summary, these data suggest that maintenance chemotherapy is associated with superior time to progression but no survival gain. However, these randomized trials did not incorporate taxane-based chemotherapeutic regimens, the new standard of care in metastatic breast cancer patients these days.

In the 10 years since their initial licensing in Europe, the taxanes, paclitaxel and docetaxel, have emerged as critical drugs in the treatment of metastatic breast cancer patients. In TAX 303 trial, patients with prior alkylating agent exposure were randomly assigned to receive either docetaxel, 100 mg/m2, or doxorubicin, 75 mg/m2, every 3 weeks. Docetaxel produced a superior response rate (48% versus 33%, P=.008) and time to treatment failure. In addition, docetaxel was less marrow suppressive, with statistically significantly lower rates of thrombocytopenia, anemia, transfusions of blood and platelets, and neutropenic fever. Paclitaxel has been compared with doxorubicin in two randomized trials. In a European Organization for Research and Treatment of Cancer study, paclitaxel (200mg/m2 administered in a 3-hour infusion) was inferior to doxorubicin . In an Eastern Cooperative Oncology Group (ECOG) trial, 24-hour paclitaxel and doxorubicin produced equivalent results . Paclitaxel has also been shown to be equivalent to CMFP (cyclophosphamide, methotrexate, fluorouracil, prednisone) chemotherapy as first-line chemotherapy for metastatic breast cancer patients .

The survival advantage of combination chemotherapy has not been firmly established in breast cancer patients yet. No trial has shown a convincing survival advantage from combination therapy over single agents given in sequence. However, all published trials have been criticized for being underpowered and unable to demonstrate survival differences as high as 20% . A 1998 metaanalysis of 1,986 patients randomly assigned between combination chemotherapy and single-agent therapy in metastatic breast cancer patients demonstrated a survival advantage to combination chemotherapy, with a hazard ratio of 0.82 (range, 0.75 to 0.90). Two recently published studies, capecitabine and docetaxel versus docetaxel alone and paclitaxel and gemcitabine versus paclitaxel alone , have shown significant survival advantages of combination chemotherapy.

In the capecitabine/docetaxel study, 511 patients with measurable metastatic breast cancer who had received a prior anthracycline were randomly assigned to receive either docetaxel and oral capecitabine or docetaxel alone [16]. The combination of docetaxel and capecitabine demonstrated a higher response rate (42% vs 30%, P=.006), longer time to progression (6.1 vs 4.2 months, P=.0001), and longer overall survival (14.5 vs 11.5 months, P=.0126). The gemcitabine/paclitaxel study randomized 529 women with chemo-naïve, measurable metastatic breast cancer to receive either paclitaxel (175 mg/m2 over 3 hours every 3 weeks) and gemcitabine (1,250 mg/m2 over 30 minutes, on days 1 and 8 every 3 weeks), or paclitaxel (175 mg/m2 over 3 hours every 3 weeks) alone. The combination arm showed higher response rates (41% vs 22%, P<.0001), longer time to progression (5.2 vs 2.9 months, P<.0001), and longer survival (18.5 vs 15.8 months, P=.018).

At the ASCO meeting 2005, Chan and colleagues reported the results of a European phase III study comparing gemcitabine/docetaxel versus capecitabine/docetaxel for anthracycline-pretreated metastatic breast cancer patients . 305 patients were randomized to receive gemcitabine/docetaxel over capecitabine/docetaxel and there were no significant difference in response rate, PFS, or survival between the two arms. However, gemcitabine/docetaxel had a better risk-benefit profile in terms of less drug-related discontinuation, less gastrointestinal toxicity, and less skin toxicities.

Although there are several randomized trials showing negative results for survival gain in patients who received maintenance chemotherapy, the role of maintenance chemotherapy with newer agents, such as docetaxel or paclitaxel, have not been established yet. The Italian MANTA trial has registered 451 metastatic breast cancer patients to receive induction chemotherapy with epirubicin or doxorubicin/paclitaxel and further randomized 253 responders (CR, PR, SD) to receive maintenance therapy with paclitaxel or observation . Although this trial demonstrated no difference in PFS or survival between the two arms, their metaanalysis advocated survival benefit of maintenance therapy. Since gemcitabine/paclitaxel (GP) combination chemotherapy is one of the two regimens which showed definite survival gain from a randomized trial, we plan to randomize patients who responded to six cycles of GP induction chemotherapy to receive additional maintenance GP chemotherapy until disease progression versus observation. We hypothesize that patients who receive maintenance GT chemotherapy will do better in terms of progression free survival.

ELIGIBILITY:
Inclusion Criteria

* Histologically Confirmed Metastatic, or Recurrent Breast Cancer
* Age over 18 Years
* ECOG Performance Status 0-2
* Premenopausal or Postmenopausal Breast Cancer Patients With Measurable or Non-Measurable Lesions, Who Are Candidates for Chemotherapy
* Life Expectancy ≥ 3 Months
* Patients May Have Received Prior Neoadjuvant or Adjuvant Taxane Regimen as Long as it Has Been 12 Months Since Completion of Regimen.
* Patients Either May or May Not Have a Prior Anthracycline Containing Regimen.
* Prior Hormonal Therapy as a Treatment of Metastatic Disease is Allowed. But Antitumoral Hormonal Therapy Must be Terminated Prior to Enrollment(up to the Date of Randomization)
* Prior Radiation Therapy Allowed as Long as < 25% of the Bone Marrow Has Been Treated,and the Patients Must Have Recovered From the Acute Toxic Effects of the Treatment Prior to Study Enrollment.Prior Radiation to the Whole Pelvis is Not Allowed. Prior Radiotherapy Must be Completed 4 Weeks Before Study Entry.
* Adequate Bone Marrow Function (≥ ANC 1,500/ul, ≥ Platelet 100,000/ul, ≥ Hemoglobin 9.0 g/dl)
* Adequate Renal Function (≤ Serum Creatinine 1.5 mg/dl or CCr ≥ 50 ml/Min)
* Adequate Liver Function (≤ Serum Bilirubin 1.5 mg/dl, ≤ AST/ALT x 3 Upper Normal Limit)
* No Prior History of Chemotherapy for Metastatic, Recurrent Breast Cancer
* Written Informed consent.

Exclusion Criteria

* Serious Uncontrolled Intercurrent Infections
* Serious Intercurrent Medical or Psychiatric Illness, Including Active Cardiac Disease
* Pregnancy or Breast Feeding
* Second Primary Malignancy(Except Cancer of Cervix or Skin or Other Malignancy Treated at Least 5 Years Previously With no Evidence of Recurrence)
* Documented Parenchymal or Leptomeningeal Brain Metastasis
* Peripheral Neuropathy ≥ Grade 2
* Prior Treatment With Gemcitabine Will Not be Allowed.
* HER-2 Overexpressing Breast Cancer and Concomitant Trastuzumab Treatment is Not Allowed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326 (Actual)
Dates: Start 2007-05; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Progression free survival | approximately 4 years

SECONDARY OUTCOMES:
a) overall survival b) quality of life c) toxicity of GP chemotherapy d) duration of response | approximately 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Young-Hyuck Im, M.D., Ph.D, Principal Investigator — Samsung Medical Center
Locations (15):
- South Korea (15):
  - Ajou University University Hospital, Suwon, Gyeonggi-do
  - Hanlym University Hospital, Anyang, Kyeongki-Do
  - Bundang Seoul National University Hospital, Bundang, Kyeongki-Do
  - Yeungnam University Hospital, Kyungsan, Kyungsangbuk-Do
  - Daegu Patima Hospital, Daegu
  - Inha University School of Medicine, Inchon
  - Seoul National University Hospital, Seoul
  - Yonsei University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - National Cancer Center, Seoul
  - Kunkuk University Hospital, Seoul
  - Ewha University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Soonchunhyang University Hospital, Seoul
  - Ulsan University Hospital, Ulsan

REFERENCES:
- [Derived] Park YH, Jung KH, Im SA, Sohn JH, Ro J, Ahn JH, Kim SB, Nam BH, Oh DY, Han SW, Lee S, Park IH, Lee KS, Kim JH, Kang SY, Lee MH, Park HS, Ahn JS, Im YH. Phase III, multicenter, randomized trial of maintenance chemotherapy versus observation in patients with metastatic breast cancer after achieving disease control with six cycles of gemcitabine plus paclitaxel as first-line chemotherapy: KCSG-BR07-02. J Clin Oncol. 2013 May 10;31(14):1732-9. doi: 10.1200/JCO.2012.45.2490. Epub 2013 Apr 8. PMID 23569309